CLINICAL TRIAL: NCT02057822
Title: Cytokine Assay in Tears of Healthy Children and With Vernal Keratocunjonctivitis: Case Control Study and Monitoring of Cases at 6 Months
Brief Title: Cytokine Assay in Tears of Healthy Children and With Vernal Keratoconjunctivitis: Case Control Study and Monitoring of Cases at 6 Months
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0170; 2012-A00034-39
Record Dates: First submitted 2013-11-25; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Vernal Keratoconjunctivitis; Healthy Children
Keywords: Vernal keratoconjunctivitis; Cytokines; Mediators; Tears
MeSH Terms: conditions — Conjunctivitis, Allergic; Lacerations

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- vernal keratoconjunctivitis: The main objective of our study was to compare the concentration of 40 cytokines in vernal keratoconjonctivitis and in control subjects
  Interventions: Procedure: Cytokins assay in tears
- healthy children: The main objective of our study was to compare the concentration of 40 cytokines in vernal keratoconjunctivitis and in control subjects
  Interventions: Procedure: Cytokins assay in tears

INTERVENTIONS:
Procedure: Cytokins assay in tears

SUMMARY:
The ocular surface may be the seat of an inflammatory process in many pathology as vernal keratoconjunctivitis. It has been shown that inflammatory cytokines produced by the cells themselves and the constituent cells of the target organ, are the main factors that cause inflammation. The main objective of our study was to compare the concentration of 40 cytokines in vernal keratoconjunctivitis and in control subjects.

DETAILED DESCRIPTION:
The ocular surface may be the seat of an inflammatory process in many pathology as vernal keratoconjunctivitis. It has been shown that inflammatory cytokines produced by the cells themselves and the constituent cells of the target organ, are the main factors that cause inflammation. The main objective of our study was to compare the concentration of 40 cytokines in vernal keratoconjunctivitis and in control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Childrens between 3 and 18 years
* Affiliated at system of French social security
* Signed by the holders of parental authority of the sheet and written consent to participate in this study
* First consultation at Clermont-Ferrand Hospital for vernal keratocunjunctivitis

Exclusion Criteria:

* Subject suffering from acute or chronic eye disease in which the physician investigator resound with the results: uveitis, glaucoma, retinopathy
* Subject who had undergone eye surgery
* Subject having an infection the day of collection: ENT, digestive, urinary
* Subject with cancer, mental illness or any other condition in which the physician investigator sound informed consent and / or the results
* Pregnant subject
* Subject with contact lenses
* Subject who judged by the investigating physician not enough cooperating to allow a safe collection

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: healthy children children with vernal keratoconjunctivitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of 40 cytokines in tears | at time 0
  Comparaison of concentration of 40 cytokines in tears between healthy children and children with vernal keratoconjunctivitis

SECONDARY OUTCOMES:
Validation of normal range of cytokines in tears of healthy children | at 6 month
Modification of the inflammatory profile according to the clinical severity and treatment | at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric CHIAMBARETTA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France